CLINICAL TRIAL: NCT03267225
Title: Study on the Genetic Determinants of Clindamycin/Rifampin Interaction
Brief Title: Genetic Determinants of Clindamycin/Rifampin Interaction
Acronym: CLINDA-RIFAM
Status: Completed | Type: Observational
Sponsor: Dr Valerie ZELLER (Other)
Collaborators: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor-Investigator, Dr Valerie ZELLER, MD, principal investigator, Groupe Hospitalier Diaconesses Croix Saint-Simon
Organization: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Other Study IDs: D-VZR_2015_3
Record Dates: First submitted 2016-09-09; First posted 2017-08-30 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: VA Drug Interaction
Keywords: drug interaction; genetic polymorphism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Main objective- To study the influence of the polymorphisms of nuclear receptor proteins pregnane X receptor (PXR), Liver X receptor alpha (LXRα), and Cytochrome P450 (CYP450) on the clindamycin clearance during clindamycin/rifampin combination therapy.

Secondary objectives To study the influence of these polymorphisms on clindamycin clearance, before combination therapy with rifampin (clindamycin monotherapy) To study the influence of these polymorphisms on CYP450 activity before combination therapy with rifampin (clindamycin monotherapy) To study the influence of these polymorphisms on the increase of CYP450 activity after clindamycin/rifampin combination therapy To study the difference between the expected and observed clindamycin serum concentrations after dosage adjustment, in patients with clindamycin dosage adjustment after combination therapy with rifampin

DETAILED DESCRIPTION:
Eligible patients will be informed on the study during their hospitalisation in the unit for the treatment of bone and joint infection by the medical doctor. If they agree to participate in the study, the following samples will be performed :

* After at least 24 hours of clindamycin therapy and before combination therapy with rifampin:

  * 1 urine sample (5 mL) for CYP 450 activity phenotyping
  * 1 blood sample (5 mL on ethylenediaminetetraacetic acid (EDTA) tubes) for measuring clindamycin serum concentration and genotyping
* After ten days of clindamycin-rifampin combination therapy:

  * 1 urine sample (5 mL) for CYP 450 activity phenotyping
  * 1 blood sample (5 mL on EDTA tubes) for measuring clindamycin serum concentration and genotyping

ELIGIBILITY:
Inclusion Criteria:

* bone or joint infection
* aged ≥ 18 years old
* treatment with clindamycin/rifampin combination therapy > 10 days

Exclusion Criteria:

* prescription of another treatment with potential action on CYP450
* pregnant or breast feeding patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient treated for a bone or joint infection with a clindamycin/rifampin combination therapy, for at least 10 days
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
Genetic polymorphism of PXR, LXRalpha, CYP450 on clindamycin clearance with clindamycin/rifampin combination therapy | 10 days after onset of clindamycin/rifampin combination therapy
  Impact of PXR, LXRα, CYP 450 3A4/A5 polymorphism on clindamycin clearance after combination clindamycin-rifampin therapy will be analyzed by studying the association of these polymorphisms and clindamycin serum concentrations.

SECONDARY OUTCOMES:
Genetic polymorphism of PXR, LXRalpha, CYP450 on clindamycin clearance before combination therapy with rifampin (clindamycin monotherapy) | One to four days after onset of clindamycin therapy and before starting rifampin therapy
  Impact of PXR, LXRα, CYP 450 3A4/A5 polymorphism on clindamycin clearance before rifampin therapy will be analyzed by studying the association of these polymorphisms and clindamycin serum concentrations.
Genetic polymorphism of PXR, LXRalpha, CYP450 on the increase of CYP 3A4 activity before combination therapy with rifampin | One to four days after onset of clindamycin therapy and before starting rifampin therapy
  Impact of PXR, LXRα, CYP 450 3A4/A5 polymorphism on CYP 450 3A activity before combination therapy with rifampin will be analyzed by studying the association of these polymorphisms and clindamycin serum concentrations.
Genetic polymorphism of PXR, LXRalpha, CYP450 on the increase of CYP 3A4 activity after clindamycin/rifampin combination therapy | 10 days after onset of clindamycin/rifampin combination therapy
  Impact of PXR, LXRα, CYP 450 3A4/A5 polymorphism on CYP 450 3A activity after combination with rifampin therapy will be analyzed by studying the association of these polymorphisms and clindamycin serum concentrations.
Difference between expected and observed clindamycine serum concentration after dosage adjustment, in patients after combination therapy with clindamycin and rifampin,. | 10 days after onset of clindamycin/rifampin combination therapy
  The gap between the predicted and observed clindamycin serum concentrations will be quantified by MPE (Mean Prediction Errors) and RMSE (Root Mean Square Prediction Errors). Dosage adjustment will be considered predictive of the concentration if MPE and RMSE are < 20 %.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Zeller, MD, Principal Investigator — GH Diaconesses Croix Saint Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, France

IPD SHARING:
Plan to Share IPD: No